CLINICAL TRIAL: NCT00604032
Title: Clinical Evaluation of the Phototoxic Potential of Atralin (Tretinoin) Gel, 0.05%
Brief Title: Study to Determine the Phototoxity of Atralin (Tretinoin) Gel, 0.05%
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Coria Laboratories, Ltd. (Industry)
Responsible Party: D. Cargill, PhD, Coria Laboratories, Ltd.
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 029-066-09-001
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-02

CONDITIONS: Healthy
Keywords: Safety when exposed to sunlight
MeSH Terms: interventions — Tretinoin; Gels

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Placebo Comparator)
  Interventions: Drug: Atralin (tretinoin) Gel, 0.05%

INTERVENTIONS:
Drug: Atralin (tretinoin) Gel, 0.05% — Assess potential of tretinoin gel, 0.05% to produce phototoxic reactions, measured 24 and 48 hours after UV radiation of drug on the skin.

SUMMARY:
To assess the potential of tretnoin gel 0.05% to produce phototoxic reactions, measured as skin reactions 24 and 48 hours after UV radiation of drug on skin.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy volunteers
* 18 years of age or older

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-01; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
UV induced skin sensitization | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Stanfiled, MS, Principal Investigator — Suncare Laboratories
Locations (1):
- Suncare Research Laboratories, Winston-Salem, North Carolina, United States